CLINICAL TRIAL: NCT01053455
Title: Observational Crossover Study Comparing Oxygenation and Ventilation Using Biphasic CPAP (SiPAP) Versus CPAP to Treat Respiratory Distress in Low Birth Weight Infants
Brief Title: Observational Crossover Study Comparing Oxygenation and Ventilation Using SiPAP Versus CPAP in LBW Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Andrea Lampland, Neonatologist, Children's Hospitals and Clinics of Minnesota
Other Study IDs: 0911-106
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Ventilation; Respiratory Distress Syndrome
Keywords: Non-invasive ventilation; SiPAP; CPAP; low birth weight infants; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Starting on NCPAP: randomized to start on NCPAP
  Interventions: Device: SiPAP
- Starting on SiPAP: randomized to SiPAP
  Interventions: Device: SiPAP

INTERVENTIONS:
Device: SiPAP — biphasic CPAP (SiPAP) to be alternated in 1 hour blocks with NCPAP

SUMMARY:
Investigation of effects of SiPAP versus NCPAP on oxygenation and ventilation in LBW infants with respiratory distress. Our hypothesis is that the LBW infants will achieve the same level of oxygenation and improved ventilation when being treated with SiPAP as compared to NCPAP.

ELIGIBILITY:
Inclusion Criteria:

1. LBW infant (birth weight <2500 grams)
2. Currently on nasal CPAP
3. Use of nasal CPAP for >24 hours prior to study initiation
4. If history of intubation with mechanical ventilation, patient will be extubated >24 hours prior to study initiation
5. FiO2 requirement of 25-50%

Exclusion Criteria:

1. FiO2 requirement >0.5
2. Congenital defects/deformities of the head, pulmonary or cardiovascular systems
3. Chromosomal abnormalities/genetic syndromes
4. Active medical treatment for symptomatic PDA
5. Active medical treatment for culture proven sepsis
6. Within 24 hours of invasive surgical procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: low birth weight infants
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lampland, MD, Principal Investigator — Childrens Hospitals and Clinics of MN - St. Paul
Locations (1):
- Childrens Hospital and Clinics of MN - St. Paul, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Lampland AL, Plumm B, Worwa C, Meyers P, Mammel MC. Bi-level CPAP does not improve gas exchange when compared with conventional CPAP for the treatment of neonates recovering from respiratory distress syndrome. Arch Dis Child Fetal Neonatal Ed. 2015 Jan;100(1):F31-4. doi: 10.1136/fetalneonatal-2013-305665. Epub 2014 Aug 1. PMID 25085943